CLINICAL TRIAL: NCT04509674
Title: EMPACT-MI: A Streamlined, Multicentre, Randomised, Parallel Group, Double-blind Placebo-controlled Superiority Trial to Evaluate the Effect of EMPAgliflozin on Hospitalisation for Heart Failure and Mortality in Patients With aCuTe Myocardial Infarction
Brief Title: EMPACT-MI: A Study to Test Whether Empagliflozin Can Lower the Risk of Heart Failure and Death in People Who Had a Heart Attack (Myocardial Infarction)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1245-0202; 2019-001037-13 (EudraCT Number)
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded investigator review of events in place of centralized adjudication.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Empagliflozin 10 mg (Experimental)
  Interventions: Drug: Empagliflozin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin
  Arms: Empagliflozin 10 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a study in adults who had a heart attack (myocardial infarction). The purpose of this study is to find out whether a medicine called empagliflozin helps to lower the chances of having to go to the hospital for heart failure and whether it lowers the chances of dying from cardiovascular disease.

People who are in hospital may join the study soon after being treated for their heart attack. Participants are put into 2 groups by chance. One group takes 1 empagliflozin tablet a day. The other group takes 1 placebo tablet a day. Placebo tablets look like empagliflozin tablets but do not contain any medicine. All participants continue their standard treatment. Empagliflozin belongs to a class of medicines known as SGLT-2 inhibitors. Empagliflozin is a medicine that helps people with type 2 diabetes to lower their blood sugar. Researchers think that empagliflozin might also help people after heart attack who are at risk for heart failure, whether or not they have diabetes.

Participants are in the study for about 1 to 2 years. During this time, there are about 4 visits inperson, 2 visits are done either by phone or by use of an mobile application. Results between the empagliflozin and placebo groups are compared. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Of full age of consent (according to local legislation, at least ≥ 18 years) at screening.
2. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
3. Male or female patients. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
4. Diagnosis of spontaneous Acute Myocardial Infarction (AMI): ST-Elevation Myocardial Infarction (STEMI) or Non-ST Elevation Myocardial Infarction (NSTEMI) with randomisation to occur no later than 14 calendar days after hospital admission. For patients with an in-hospital Myocardial Infarction (MI) as qualifying event, randomization must still occur within 14 days of hospital admission.
5. High risk of HF, defined as EITHER

   1. Symptoms (e.g. dyspnea; decreased exercise tolerance; fatigue), or signs of congestion (e.g. pulmonary rales, crackles or crepitations; elevated jugular venous pressure; congestion on chest X-ray), that require treatment (e.g. augmentation or initiation of oral diuretic therapy; i.v. diuretic therapy; i.v. vasoactive agent; mechanical intervention etc.) at any time during the hospitalization.

      OR
   2. Newly developed Left Ventricular Ejection Fraction (LVEF) < 45% as measured by echocardiography, ventriculography, cardiac Computer Tomography (CT), Magnetic Resonance Imaging (MRI) or radionuclide imaging during index hospitalisation.
6. In addition at least one of the following risk factors:

   * Age > 65 years,
   * Newly developed LVEF < 35%,
   * Prior MI (before index MI) documented in medical records,
   * Estimated Glomerular Filtration Rate (eGFR) < 60 ml/min/1.73m2 (using Chronic Kidney Disease Epidemiology Collaboration Equation (CKD-EPI) formula based on creatinine from local lab at any time during index hospitalisation),
   * Atrial fibrillation (persistent or permanent ; if paroxysmal, only valid if associated with index MI),
   * Type 2 diabetes mellitus (prior or new diagnosis),
   * N-Terminal Pro-Brain Natriuretic Peptide (NT-proBNP) >1,400 pg/mL for patients in sinus rhythm, >2,800 pg/mL if atrial fibrillation; Brain Natriuretic Peptide (BNP) >350 pg/mL for patients in sinus rhythm, >700 pg/mL if atrial fibrillation, measured at any time during hospitalisation,
   * Uric acid >7.5 mg/dL (>446 μmol/L), measured at any time during hospitalisation,
   * Pulmonary Artery Systolic Pressure [or right ventricular systolic pressure] >40 mmHg (non-invasive [usually obtained from clinically indicated post-MI echocardiography] or invasive, at any time during hospitalisation),
   * Patient not revascularized (and no planned revascularization) for the index MI (Includes e.g. patients where no angiography is performed, unsuccessful revascularization attempts, diffuse atherosclerosis not amenable for intervention; but does NOT include if revascularization was not performed due to nonobstructive coronary arteries),
   * 3-vessel coronary artery disease at time of index MI,
   * Diagnosis of peripheral artery disease (extracoronary vascular disease, e.g. lower extremity artery disease or carotid artery disease).

Exclusion Criteria:

1. Diagnosis of chronic Heart Failure (HF) prior to index MI.
2. Systolic blood pressure < 90 mmHg at randomisation.
3. Cardiogenic shock or use of i.v. inotropes in last 24 hours before randomisation.
4. Coronary Artery Bypass Grafting planned at time of randomisation.
5. Current diagnosis of Takotsubo cardiomyopathy.
6. Any current severe (stenotic or regurgitant) valvular heart disease.
7. eGFR < 20 ml/min/1.73m2 (using CKD-EPI formula based on most recent creatinine from local lab during index hospitalisation) or on dialysis.
8. Type I diabetes mellitus. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6522 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2023-11-05 (Actual); Study Completion 2023-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (436):
- United States (85):
  - Advanced Cardiovascular LLC, Alexander City, Alabama
  - Grandview Medical Center, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Arkansas Cardiology, PA, Little Rock, Arkansas
  - Comprehensive Cardiovascular Medical Group, Bakersfield, California
  - Valley Clinical Trials, Inc., Covina, California
  - Cardiovascular Innovation and Research Center, Long Beach, California
  - University of California Los Angeles, Los Angeles, California
  - InvivoCure, Mission Hills, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Valley Clinical Trials, Inc., Pasadena, California
  - Kaiser Permanente, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Interventional Cardiology Medical Group, West Hills, California
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Integrative Research Associates, Fort Lauderdale, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Cardiology Partners Clinical Research Institute, Palm Beach Gardens, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Cardiovascular Consultants of South Georgia, LLC, Thomasville, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - Advanced Heart Care, LLC, Medicoricum, LLC, Fairview Heights, Illinois
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Cardiovascular Specialists of Central Maryland, Columbia, Maryland
  - Shady Grove Adventist Hospital, Rockville, Maryland
  - Healthy Heart Cardiology, Grand Rapids, Michigan
  - Western Michigan University, Kalamazoo, Michigan
  - Mid Michigan Medical Center, Midland, Michigan
  - Michigan Heart, PC, Ypsilanti, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Missouri Cardiovascular Specialists, LLP, Columbia, Missouri
  - University of Missouri Health System, Columbia, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Gateway Cardiology, PC, St Louis, Missouri
  - St. Louis Heart and Vascular, P.C., St Louis, Missouri
  - Holy Name Medical Center, Hackensack, New Jersey
  - AtlantiCare, Pomona, New Jersey
  - The Heart House, Vineland, New Jersey
  - SJH Cardiology Associates, Liverpool, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moses H. Cone Memorial Hospital, Greensboro, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - North Carolina Heart and Vascular, Raleigh, North Carolina
  - Trinity Health Center Medical Arts, Minot, North Dakota
  - Aultman Hospital, Canton, Ohio
  - Cincinnati VA Medical Center, Cincinnati, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Oklahoma Heart Hospital Research Foundation, Incorporated, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research Group, Oklahoma City, Oklahoma
  - Capital Area Research, LLC, Camp Hill, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Guthrie Medical Group PC, Sayre, Pennsylvania
  - Upstate Cardiology, PA, Greenville, South Carolina
  - Carolina Heart Specialists, LLC, Lancaster, South Carolina
  - Monument Health, Rapid City, South Dakota
  - Centennial Heart Cardiovascular Consultants, LLC, Nashville, Tennessee
  - Parkway Cardiology Associates, Oak Ridge, Tennessee
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - Texas Health Presbyterian Hospital Allen, Allen, Texas
  - Amarillo Heart Clinical Research Institute, Incorporated, Amarillo, Texas
  - Pharmatex Research, Amarillo, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Baylor Scott and White Health, Plano, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Revival Research Institute, LLC., Sherman, Texas
  - Cardiovascular Associates of East Texas, PA, Tyler, Texas
  - Carient Heart and Vascular, Manassas, Virginia
  - Riverside Regional Medical Center, Newport News, Virginia
  - Tidewater Physicians Multispecialty Group, Newport News, Virginia
  - Sentara Hospitals, Norfolk, Virginia
  - Roanoke Heart Institute PLC, Roanoke, Virginia
- Argentina (20):
  - Instituto Cardiovascular de Buenos Aires, Belgrano
  - Fundacion Sanatorio Güemes, Ciudad Autonoma Buenos Aires
  - Centro de Investigacion Clinica Coronel Suarez, Coronel Suárez
  - Instituto de Cardiologia de Corrientes, Corrientes
  - Hospital Italiano de Córdoba, Córdoba
  - Sanatorio Allende, Córdoba
  - Centro Medico Luquez, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Clinica Privada del Prado, Córdoba
  - Fundación Favaloro para la Docencia e Investigación Medica, Montserrat
  - Sanatorio Modelo de Quilmes, Quilmes
  - Instituto Cardiovascular de Rosario, Rosario
  - Sanatorio Delta, Rosario
  - Sanatorio Parque, Rosario
  - Corporacion Medica de Gral. San Martin S.A., San Martín
  - Centro Privado de Cardiologia, San Miguel de Tucumán
  - Clinica U.O.M., San Nicolás
  - Sanatorio Diagnóstico, Santa Fe
  - Hospital "Dr. José Maria Cullen", Santa Fé
  - Clinica Privada Fusavim SRL, Villa María
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - South Western Sydney Local Health District, Liverpool, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Alfred Hospital, Melbourne, Victoria
- Brazil (26):
  - JMF Clinica Do Coracao LTDA, Aracaju - SE
  - Hospital Santa Isabel, Balneário Camboriú
  - Hospital Madre Teresa, Belo Horizonte
  - Hospital do Coracao do Brasil, Brasília
  - Hospital Angelina Caron, Campina Grande do Sul
  - Centro Especializado em Cardiol Loema Instituto de Pesq Clin, Campinas
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas
  - Hospital de Messejana Dr. Carlos Alberto Studart Gomes, Fortaleza
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia
  - Hospital Regional Hans Dieter Schmidt, Joinville
  - Santa Casa de Misericórdia de Marília, Marília
  - Hospital São Vicente de Paulo, Passo Fundo
  - Hospital Sao Lucas da PUCRS, Porto Alegre
  - Instituto de Cardiologia Rio Grande do Sul, Porto Alegre
  - Hospital Nossa Senhora da Conceição, Porto Alegre
  - Hospital Agamenon Magalhaes, Recife
  - Fundacao de apoio ao ensino e assitencia HCFMRP, Ribeirão Preto
  - Hospital Copa D'or, Rio de Janeiro
  - Instituto de Ensino E Pesquisa Do Hospital Da Bahia, Salvador
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Hospital de Base - Fac Med de Sao Jose do Rio Preto, São José do Rio Preto
  - Hospital Samaritano, São Paulo
  - Hospital Sao Luiz Jabaquara, São Paulo
  - Hospital Sao Luiz Morumbi, São Paulo
  - Hospital das Clínicas de Sao Paulo - INCOR, São Paulo
  - Santa Casa de Votuporanga, Votuporanga
- Bulgaria (17):
  - Multiprofile Hospital For Active Treatment Pulse AD, Blagoevgrad
  - Multiprofile Hospital For Active Treatment "Dr. Tota Venkova" AD, Gabrovo
  - Multiprofile Hospital for Active Treatment AD Haskovo, Haskovo
  - Multiprofile Hospital For Active Treatment - Pazardzhik AD, Pazardzhik
  - Specialized Hospital for Active Treatment Sv. Georgi - Pernik, Pernik
  - Medical Center Medconsult Pleven LTD, Pleven
  - Multiprofile Hospital for Active Treatment Heart and Brain EAD, Pleven
  - SHAT in Cardiology EAD, Pleven, Pleven
  - Hospital MHAT Plovdiv, AD, Plovdiv
  - National Heart Hospital, Sofia, Sofia
  - City Clin.Univ.MPHAT EOOD,Clin.of Cardiology, Sofia, Sofia
  - University Multiprofile Hospital for Active Treatement "Alexandrovska" EAD, Sofia
  - UMHAT "Tsaritsa Yoannalsul", Sofia
  - Medical Military Academy MHAT Sofia, Sofia
  - Multiprofile Hospital MHATEM 'Pirogov', Sofia, Sofia
  - MHAT Sv.Anna, Clinic of Internal Diseases, Sofia, Sofia
  - Hospital Trakia Park, Stara Zagora
- Canada (27):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Royal Inland Hospital, Kamloops, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - GA Research Associates Ltd., Moncton, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - William Osler Health Centre, Brampton, Ontario
  - Queen's University, Kingston, Ontario
  - One Heart Care Ventures, Mississauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Peterborough Regional Health Centre, Peterborough, Ontario
  - Heart Health Institute, Scarborough Village, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - IUCPQ (Laval University), Sainte-Foy, Quebec
  - CIUSSS de l Estrie-CHUS, Sherbrooke, Quebec
  - CSSS du Sud de Lanaudiere - Hopital Pierre-Le Gardeur, Terrebonne (Lachenaie), Quebec
  - CIUSSS de la Mauricie-et-du-Centre-du-Quebec, Trois-Rivières, Quebec
  - Prairie Vascular Research Inc., Regina, Saskatchewan
  - Oakville Trafalgar Memorial Hospital, Oakville
- China (19):
  - Beijing Chao-Yang Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Beijing Luhe Hospital Capital Medical University, Beijing
  - Changsha Central Hospital, Changsha
  - Xiangya Hospital, Central South University, Changsha
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital of Harbin Medical University, Haerbin
  - Hainan General Hospital, Haikou
  - Shulan(Hanghzhou) Hospital, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - The Second Affiliated Hospital of Lanzhou Medical University, Lanzhou
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - People's Hospital of Liaoning Province, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Renmin Hospital of Wuhan University, Wuhan
- Denmark (6):
  - Aalborg Universitetsshospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Frederiksberg Hospital, Frederiksberg
  - Herlev and Gentofte Hospital, Herlev
  - Slagelse Sygehus, Slagelse
- France (8):
  - HOP Sud Francilien, Corbeil-Essonnes
  - HOP CHU de Grenoble, Grenoble
  - CHRU Lille, Lille
  - Hospital de Saint Joseph et Saint Luc, Lyon
  - HOP Bichat, Paris
  - CHU Rouen, Rouen
  - HOP Trousseau, Tours
  - HOP Brabois, Vandœuvre-lès-Nancy
- Germany (19):
  - SLK-Kliniken Heilbronn GmbH, Bad Friedrichshall
  - Kerckhoff-Klinik, Bad Nauheim, Bad Nauheim
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn AöR, Bonn
  - Bremer Institut für Herz- und Kreislaufforschung (BIHKF) am Klinikum Links der Weser, Bremen
  - Klinikum Coburg gGmbH, Coburg
  - St. Johannes Hospital Dortmund, Dortmund
  - Städtisches Klinikum Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main
  - Universitäts-Herzzentrum Freiburg, Bad Krozingen GmbH, Freiburg I. Breisgau
  - Asklepios Kliniken GmbH & Co. KGaA, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Ambulantes Herzzentrum Kassel, Kassel
  - Universitätsklinikum Leipzig, Leipzig
  - Katholisches Klinikum Mainz, Mainz
  - Clemenshospital, Münster
  - Kardiologische Praxis Papenburg, Papenburg
  - Universitätsklinikum Regensburg, Regensburg
- Hungary (15):
  - Lausmed Kft. Outpatient Unit of Internal Medicine, Baja
  - Buda Hospital of the Hospitaller Order of Saint John of God, Budapest
  - Semmelweis University, Budapest
  - St. Imre Hospital, Budapest, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Jahn Ferenc Del-Pest Hospital, Budapest
  - University Debrecen Hospital, Debrecen
  - Csongrad Megyei Eu. Ellato Kozp. Hodmezovasarhely-Mako, Hódmezővásárhely
  - Somogy County Kaposi Mor Teaching Hospital, Kaposvár
  - Bacs-Kiskun Megyei Onkormanyzat Hospital, Kecskemét
  - Pest Megyei Flor Ferenc Hospital, Kistarcsa
  - University of Szeged, Szeged
  - Fejer County Saint George University Teaching Hospital, Székesfehérvár
  - Jasz-Nagykun-Szolnok Megyei Hetenyi G. Korhaz-Rendelointezet, Szolnok
  - Zala County Hospital, Zalaegerszeg, Zalaegerszeg
- India (13):
  - Kamalnayan Bajaj Hospital, Aurangabad
  - Sri Jayadeva Institute of Cardiovascular Sciences & Research, Bangalore
  - Narayana Institute of Cardiac Sciences, Bangalore
  - KLES Dr.Prabhakar Kore Hospital and Medical Research Centre, Belagavi
  - Madras Medical Mission,, Chennai
  - Eternal Heart Care Centre & Research Institute Pvt. Ltd., Jaipur
  - KEM Hospital and Seth G S Medical College, Mumbai
  - Sion Hospital (Lokmanya Tilak Municipal Hospital), Mumbai
  - Government Medical College & Hospital, Nagpur
  - GB Pant Institute of Post Graduate Medical Education and Research, New Delhi
  - Max Superspeciality Hospital, New Delhi
  - Sir Gangaram Hospital, New Delhi
  - Sahyadri Speciality Hospital, Pune
- Israel (19):
  - Haemek Medical Center, Afula
  - Assuta Medical Center, Ashdod
  - Barzilai Medical Center, Ashkelon
  - Assaf Harofe Medical Center, Beer Yaacov
  - Soroka Univ. Medical Center, Beersheba
  - Hillel Yaffe Medical Center, Hadera, Hadera
  - Rambam Medical Center, Haifa
  - Bnei Zion Medical Center, Haifa, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem
  - Meir Medical Center, Kfar Saba
  - West.Galilee Med.Cent.Naharia, Nahariya
  - Rabin Medical Center Beilinson, Petah Tikva
  - The Chaim Sheba Medical Center Tel HaShomer, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Sourasky Medical Center, Tel Aviv
  - Baruch Padeh Medical Center, Tiberias
- Japan (29):
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - Toyota Memorial Hospital, Aichi, Toyota
  - Chibanishi General Hospital, Chiba, Matsudo
  - Seikeikai New Tokyo Heart Clinic, Chiba, Matsudo
  - Saiseikai Fukuoka General Hospital, Fukuoka, Fukuoka
  - Gifu Prefectural General Medical Center, Gifu, Gifu
  - Ogaki Municipal Hospital, Gifu, Ogaki
  - Hiroshima General Hospital, Hatsukaichi
  - Hiroshima Prefectural Hospital, Hiroshima, Hiroshima
  - Hyogo Brain and Heart Center, Hyogo, Himeji
  - Ibaraki Prefectural Central Hospital, Ibaraki, Kasama
  - Tsuchiura Kyodo General Hospital, Ibaraki, Tsuchiura
  - Ishikawa Prefectural Central Hospital, Ishikawa, Kanazawa
  - Juntendo University Shizuoka Hospital, Izunokuni
  - Tokai University Hospital, Kanagawa, Isehara
  - Sagamihara Kyodo Hospital, Kanagawa, Sagamihara
  - Yokohama City University Medical Center, Kanagawa, Yokohama
  - Fukuoka Tokushukai Hospital, Kasuga
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto, Kumamoto
  - Kusatsu General Hospital, Kusatsu
  - Miyazaki Medical Association Hospital, Miyazaki
  - Nagano Chuo Hospital, Nagano, Nagano
  - Osaka Police Hospital, Osaka, Osaka
  - Kagawa Prefectural Central Hospital, Takamatsu
  - Tokushima Prefectural Central Hospital, Tokushima
  - St. Luke's International Hospital, Tokyo, Chuo-ku
  - Tokyo Bay Urayasu Ichikawa Medical Center, Urayasu
  - Showa University Fujigaoka Hospital, Yokohama
- Netherlands (22):
  - Jeroen Bosch Ziekenhuis-Hertogenbosch, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Amsterdam UMC Locatie VUMC, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Amphia Ziekenhuis, Breda
  - IJsselland Ziekenhuis, Capelle aan den IJssel
  - Catharina Ziekenhuis, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Admiraal de Ruyter Ziekenhuis, Goes
  - Universitair Medisch Centrum Groningen, Groningen
  - Spaarne Ziekenhuis, Haarlem
  - Zuyderland Medisch Centrum, Heerlen
  - Tergooi Ziekenhuis, Hilversum
  - Vasculair Onderzoek Centrum, Hoorn
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Alrijne Ziekenhuis, Leiden
  - Ziekenhuis Rivierenland, Tiel
  - Tweesteden Ziekenhuis, locatie Tilburg, Tilburg
  - Isala Zwolle, Zwolle
- Poland (21):
  - American Heart of Poland, Bełchatów
  - Univ. Clinic Hosp, Bialystok, Bialystok
  - American Heart of Poland Sp. z o.o., Bielsko-Biala
  - American-Polish Heart Clinic, Lesser Poland Cardiovascular Centre, Chorzów
  - American Heart of Poland Sp. z o.o., Dąbrowa Górnicza
  - NZOZ Pro-Cordis Sopockie Centrum Bad. Kardiolog., Gdynia
  - Silesian Medical University in Katowice, Katowice
  - American Heart of Poland Sp. z o.o., Kędzierzyn-Koźle
  - University Hospital in Krakow, Krakow
  - The John Paul II Hosp.,Dept.of Coronary Heart Disease,Krakow, Krakow
  - Podhalanski Special.Hosp,Intern.Med&Cardiology Dept,Nowy Tag, Nowy Targ
  - Mazowiecki Szpital Specjalistyczny im. dr Jozefa Psarskiego, Ostrołęka
  - Medicome Limited Liability Company, Oświęcim
  - Independent Public Healthcare, Dept. of Cardiology, Pulawy, Puławy
  - American Heart of Poland Sp. z o.o., Sztum
  - American Heart of Poland Sp. z o.o., Tychy
  - Central Hospital of Medical Academy, Warsaw, Warsaw
  - Instytut Kardiologii, Warszawa, Warsaw
  - Dr Alfred Sokołowski Specialist Hospital, Wałbrzych
  - Jan Mikulicz-Radecki UnivClinic Hosp,Cardiology Dept,Wroclaw, Wroclaw
  - 4. Military Clinical Hospital with Polyclinic SP ZOZ, Wroclaw
- Romania (20):
  - Emergency Clinical County Hospital, Baia Mare, Baia Mare
  - Spitalul Clinic De Urgenta "Prof. Dr. Agrippa Ionescu", Baloteşti
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Spitalul Judetean de Urgenta Braila, Brăila
  - Military Central Clinical Emergency Hospital, Bucharest
  - Elias Emergency Hospital, Bucharest, Bucharest
  - Prof.C.C.Iliescu Hospital, National Institute of Cardiology, Bucharest
  - Emergency Clinical Hospital "Bagdasar-Arseni", Bucharest
  - Emergency University Hospital, Bucharest, Bucharest
  - Heart Institute "Niculae Stancioiu", Cluj Napoca, Cluj-Napoca
  - Clincal Reabilitation Hospital, Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean, Craiova, Craiova
  - Cardiovascular Diseases Institute "Prof. Georgescu", Iasi, Iași
  - SC Cardiomed SRL, Iasi, Iași
  - SC Endodigest SRL, Oradea
  - Sal Med Srl, Piteşti
  - Emergency County Clinical Hospital, Sibiu, Sibiu
  - Centrul Medical Cardiomed, Târgu Mureş
  - Country Clinical Emergency Hospital, Targu-Mures, Târgu Mureş
  - Cardiology and Cardiovascular Rehabilitation Clinic, Timișoara
- Russia (17):
  - First City Clinical Hospital named after E. E. Volosevich, Arkhangelsk
  - Regional Clinical Hospital, Kirov, Kirov
  - Regional Clinical Hospital No.1 named after Professor. S.V. Ochapovskiy, Krasnodar
  - State Healthcare Institution Clinical Hosp. No. 51, Moscow, Moscow
  - Reg.Clin.Hosp.n.a.Semashko, Nizhny Novgorod
  - Penza Regional Clinical Hospital named after N.N.Burdenko, Penza
  - Republic Kareliya Republican Hosp. named after V.A. Baranov, Petrozavodsk
  - GUZ Ryazanskiy Regional Clin. Cardiology Dispensary, Ryazan, Ryazan
  - Saint-Petersburg I.I. Dzhanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - Medical Academy named after I. Mechnikov, St. Petersburg, Saint Petersburg
  - Samara Regional Clinical Cardiology Clinic, Day Hosp. Dept., Samara
  - Saratov State Med.Univ.n.a.Razumovskogo, Saratov
  - Saratov Regional Cardiac Center, Saratov
  - Komi Republican Cardiological Dispensary, Syktyvkar
  - Regional clinical hospital, Tver, Tver'
  - Tyumen Cardiology Center, Dept.of Cardiac Arrhythmia, Tyumen
  - State Budg.Healthc.Instit Volgograd RegClin.Cardiology Centr, Volgograd
- Serbia (15):
  - Institute for Cardiovascular diseases Dedinje, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Dr. Dragisa Misovic, Belgrade
  - Clinical Medical Center Zvezdara, Belgrade, Belgrade
  - Institute of Cardiovascular Diseases, Kamenitz
  - University Clinical Center of Kragujevac, Kragujevac
  - General Hospital Leskovac, Leskovac
  - University Clinical Center Nis, Niš
  - Institute for Treatment and Rehabilitation, Niska Banja, Niška Banja
  - General Hospital Pancevo, Pančevo
  - General Hospital Sremska Mitrovica, Sremska Mitrovica
  - General Hospital Subotica, Internal Medicine, Subotica
  - Health Center Uzice, Užice
  - Health Centre Zajecar, Zaječar
  - General Hospital - Djordje Joanovic, Zrenjanin
- South Korea (7):
  - Bucheon Sejong Hospital, Bucheon-si
  - Pusan National Univ. Hosp, Busan
  - Chungbuk National University Hospital, Cheongiu
  - Chungnam National University Hospital, Daejoen
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Yonsei University Wonju Severance Christian Hospital, Wonju-si, Gangwon State
- Spain (5):
  - Hospital Germans Trias i Pujol, Badalona
  - University Hospital of Bellvitge, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari Joan XXIII, Tarragona
  - Complejo Hospitalario Universitario de Vigo, Vigo
- Ukraine (18):
  - Cherkasy Regional Cardiological Center, Cherkasy
  - City Joint Emergency Hospital, Dnepropetrovsk, Dnipro
  - Ivano-Frankivsk City Central Clinical Hospital, Ivano-Frankivsk
  - Clinical Treatment and Diagnostic Center of the Limited Liability Company "SIMEDGROUP", Ivano-Frankivsk
  - L.T. Malaya Institute of Therapy AMS of Ukraine, Kharkiv
  - Reg.Clin.Hosp.Non-Commercial Enterprise, Kharkiv
  - CI of Healthcare Kharkiv CCH #8, Kharkiv, Kharkiv
  - Khmelnytskyi Regional Hospital, Khmelnytskyi
  - Kiev City Clinical Hospital No. 5, Kiev
  - SI NSC M.D. Strazhesko Institute Cardiology of NAMSU, Kyiv, Kiev
  - City Clinical Hospital No. 1, Kiev, Kiev
  - Kiev Emergency Care Hospital, Kiev
  - Lutsk City Clinical Hospital, Lutsk
  - Communal Noncommercial Enterprise of Lviv Regional Council "Lviv Regional Clinical Psychiatric Hospital", Lviv
  - Odesa Regional Clinical Hospital, Odesa
  - Regional Clinical Hospital, Ternopil, Ternopil
  - Municipal Non-Profit Enterprise "Zakarpattia Regional Clinical Center of Cardiology and Cardiac Surgery" of Zakarpattia Regional Council, Uzhhorod
  - Zhytomyr Regional Clinical Hospital, Dept. Endocrinology, Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Udell JA, Petrie MC, Jones WS, Anker SD, Harrington J, Mattheus M, Seide S, Amir O, Bahit MC, Bauersachs J, Bayes-Genis A, Chen Y, Chopra VK, Figtree G, Ge J, Goodman SG, Gotcheva N, Goto S, Gasior T, Jamal W, Januzzi JL, Jeong MH, Lopatin Y, Lopes RD, Merkely B, Martinez-Traba M, Parikh PB, Parkhomenko A, Ponikowski P, Rossello X, Schou M, Simic D, Steg PG, Szachniewicz J, van der Meer P, Vinereanu D, Zieroth S, Brueckmann M, Sumin M, Bhatt DL, Hernandez AF, Butler J. Left Ventricular Function, Congestion, and Effect of Empagliflozin on Heart Failure Risk After Myocardial Infarction. J Am Coll Cardiol. 2024 Jun 11;83(23):2233-2246. doi: 10.1016/j.jacc.2024.03.405. Epub 2024 Apr 6. PMID 38588929
- [Derived] Butler J, Jones WS, Udell JA, Anker SD, Petrie MC, Harrington J, Mattheus M, Zwiener I, Amir O, Bahit MC, Bauersachs J, Bayes-Genis A, Chen Y, Chopra VK, Figtree G, Ge J, Goodman SG, Gotcheva N, Goto S, Gasior T, Jamal W, Januzzi JL, Jeong MH, Lopatin Y, Lopes RD, Merkely B, Parikh PB, Parkhomenko A, Ponikowski P, Rossello X, Schou M, Simic D, Steg PG, Szachniewicz J, van der Meer P, Vinereanu D, Zieroth S, Brueckmann M, Sumin M, Bhatt DL, Hernandez AF. Empagliflozin after Acute Myocardial Infarction. N Engl J Med. 2024 Apr 25;390(16):1455-1466. doi: 10.1056/NEJMoa2314051. Epub 2024 Apr 6. PMID 38587237
- [Derived] Hernandez AF, Udell JA, Jones WS, Anker SD, Petrie MC, Harrington J, Mattheus M, Seide S, Zwiener I, Amir O, Bahit MC, Bauersachs J, Bayes-Genis A, Chen Y, Chopra VK, A Figtree G, Ge J, G Goodman S, Gotcheva N, Goto S, Gasior T, Jamal W, Januzzi JL, Jeong MH, Lopatin Y, Lopes RD, Merkely B, Parikh PB, Parkhomenko A, Ponikowski P, Rossello X, Schou M, Simic D, Steg PG, Szachniewicz J, van der Meer P, Vinereanu D, Zieroth S, Brueckmann M, Sumin M, Bhatt DL, Butler J. Effect of Empagliflozin on Heart Failure Outcomes After Acute Myocardial Infarction: Insights From the EMPACT-MI Trial. Circulation. 2024 May 21;149(21):1627-1638. doi: 10.1161/CIRCULATIONAHA.124.069217. Epub 2024 Apr 6. PMID 38581389
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Streamlined, randomised, placebo-controlled, double-blind, parallel-group trial in acute myocardial infarction (MI) hospitalised patients with high-risk for subsequent hospitalization for heart failure (HHF) and mortality. Patients were randomised 1:1 to empagliflozin or placebo within 14 days of hospitalisation. Patients were treated and remained in the trial until approximately a total number of 532 patients had primary endpoint events (i.e. event driven).
Pre-assignment Details: All patients were screened for eligibility prior to participation in the trial. Patients attended a specialist site which ensured all inclusion and none of the exclusion criteria were met. Patients were not to be allocated to a treatment group if any of the entry criteria were violated. The randomised set included all randomised patients, whether treated or not. A patient randomised in error after death (i.e. mis-randomization) would be excluded as per statistical analysis plan definition.
Groups:
- Placebo: Patients with an acute myocardial infarction event took, on top of standard of care, one placebo matching-empagliflozin 10 milligrams (mg) film-coated tablet, orally, once daily, at the same time every morning, with a glass of water.
- Empagliflozin 10 mg: Patients with an acute myocardial infarction event took, on top of standard of care, one empagliflozin (Jardiance®) 10 milligrams (mg) film-coated tablet, orally, once daily, at the same time every morning, with a glass of water.
Period: Overall Study
Arm/Group | Placebo | Empagliflozin 10 mg
Started | 3262 | 3260
Treated | 3229 | 3234
Completed (Patients who did not prematurely discontinue study treatment.) | 2513 | 2550
Not Completed | 749 | 710
Not completed — Not treated | 33 | 26
Not completed — Protocol Violation | 9 | 10
Not completed — Lost to Follow-up | 31 | 39
Not completed — Patient refusal to continue, not due to adverse event | 452 | 418
Not completed — Adverse event, serious fatal event | 11 | 4
Not completed — Adverse event, non-fatal event | 107 | 118
Not completed — Other reason than listed | 106 | 95

BASELINE CHARACTERISTICS:
Population: Randomised set (RS): All randomised patients, whether treated or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empagliflozin 10 mg | Total
Number analyzed (Participants) | 3262 | 3260 | 6522
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (10.8) | 63.6 (11.0) | 63.6 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 813 | 812 | 1625
  Male | 2449 | 2448 | 4897
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 331 | 338 | 669
  Not Hispanic or Latino | 2859 | 2866 | 5725
  Unknown or Not Reported | 72 | 56 | 128
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2721 | 2730 | 5451
  Black/African-American | 48 | 44 | 92
  Asian | 413 | 421 | 834
  Other, including mixed race | 7 | 9 | 16
  Missing | 73 | 56 | 129

OUTCOME MEASURES:

1. Primary Outcome: Composite of Time to First Heart Failure Hospitalisation or All-cause Mortality
Description: The composite of time to first heart failure hospitalization or all-cause mortality is reported as the incidence rate of the first occurrence of hospitalization for heart failure (HHF) or death, whichever is earliest.
  The incidence rate was calculated as: the number of patients with an event for hospitalization for heart failure or death by treatment group during time at risk divided by the total time patients were at risk in that treatment group multiplied by 100 (per 100 Pt-years, Pt as abbreviation of patient).
Time Frame: From randomisation or first study drug administration (if randomisation occurred after first drug administration), until individual day of trial completion. Up to 1004 days.
Population: Randomised set (RS): All randomised patients, whether treated or not.
Measure: Number (95% Confidence Interval); unit: Pt with events/100 pt-years at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3262 | 3260
Pt with events/100 pt-years at risk | 6.58 [5.86 to 7.35] | 5.85 [5.17 to 6.57]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; The primary endpoint was analysed using a Cox proportional hazards model with treatment, type-2 diabetes at baseline, geographical region, age at baseline, estimated glomerular filtration rate at baseline, left ventricular ejection fraction at baseline, persistent or permanent atrial fibrillation at baseline, prior myocardial infarction at baseline, peripheral artery disease at baseline and smoking at baseline as covariates; Test type: Superiority; p = 0.2061, Regression, Cox — Null hypothesis: there is no difference regarding the risk of the endpoint in question between empagliflozin and placebo. p<=0.05 required for testing of subsequent key secondary endpoint hypotheses; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.76 to 1.06] — Empagliflozin vs. Placebo

2. Secondary Outcome: Key Secondary Endpoint - Total Number of Hospitalisations for Heart Failure (HHF) or All-cause Mortality
Description: The total number of hospitalisations for heart failure (HHF) or all-cause mortality is reported using the adjusted event rate.
  The adjusted event rate is based on a negative binomial model adjusted for treatment and type-2 diabetes at baseline, geographical region, age at baseline, estimated glomerular filtration rate at baseline, left ventricular ejection fraction at baseline, persistent or permanent atrial fibrillation at baseline, prior myocardial infarction at baseline, peripheral artery disease at baseline and smoking at baseline as covariates. The log(observation time) was used as an offset variable.
Time Frame: as for outcome 1
Population: Randomised set (RS): All randomised patients, whether treated or not.
Measure: Number (95% Confidence Interval); unit: Events/100 patient-years at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3262 | 3260
Events/100 patient-years at risk | 8.25 [6.92 to 9.83] | 7.14 [5.91 to 8.63]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — The statistical model used was a negative binomial model, including factors for treatment and type-2 diabetes at baseline, geographical region, age at baseline, estimated glomerular filtration rate at baseline, left ventricular ejection fraction at baseline, persistent or permanent atrial fibrillation at baseline, prior myocardial infarction at baseline, peripheral artery disease at baseline and smoking at baseline as covariates. The log(observation time) was used as an offset variable; p = 0.2423, Negative binomial regression; Adjusted event rate ratio = 0.87, 95% CI 2-sided [0.68 to 1.10] — Empagliflozin vs. Placebo

3. Secondary Outcome: Key Secondary Endpoint - Total Number of Non-elective Cardiovascular (CV) Hospitalisations or All-cause Mortality
Description: The total number of non-elective cardiovascular (CV) hospitalisations or all-cause mortality is reported using the adjusted event rate.
  The adjusted event rate is based on a negative binomial model adjusted for treatment and type-2 diabetes at baseline, geographical region, age at baseline, estimated glomerular filtration rate at baseline, left ventricular ejection fraction at baseline, persistent or permanent atrial fibrillation at baseline, prior myocardial infarction at baseline, peripheral artery disease at baseline and smoking at baseline as covariates. The log(observation time) was used as an offset variable.
Time Frame: as for outcome 1
Population: Randomised set (RS): All randomised patients, whether treated or not.
Measure: Number (95% Confidence Interval); unit: Events/100 patient-years at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3262 | 3260
Events/100 patient-years at risk | 16.90 [15.10 to 18.92] | 15.52 [13.82 to 17.43]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.2867, Negative binomial regression; Adjusted event rate ratio = 0.92, 95% CI 2-sided [0.78 to 1.07] — Empagliflozin vs. Placebo

4. Secondary Outcome: Key Secondary Endpoint - Total Number of Non-elective All-cause Hospitalisations or All-cause Mortality
Description: The total number of non-elective all-cause hospitalisations or all-cause mortality is reported using the adjusted event rate.
  The adjusted event rate is based on a negative binomial model adjusted for treatment and type-2 diabetes at baseline, geographical region, age at baseline, estimated glomerular filtration rate at baseline, left ventricular ejection fraction at baseline, persistent or permanent atrial fibrillation at baseline, prior myocardial infarction at baseline, peripheral artery disease at baseline and smoking at baseline as covariates. The log(observation time) was used as an offset variable.
Time Frame: as for outcome 1
Population: Randomised set (RS): All randomised patients, whether treated or not.
Measure: Number (95% Confidence Interval); unit: Events/100 patient-years at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3262 | 3260
Events/100 patient-years at risk | 26.28 [23.92 to 28.87] | 22.96 [20.84 to 25.31]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0463, Negative binomial regression; Adjusted event rate ratio = 0.87, 95% CI 2-sided [0.7654 to 0.9978] — Empagliflozin vs. Placebo

5. Secondary Outcome: Key Secondary Endpoint - Total Number of Hospitalisations for Myocardial Infarction (MI) or All-cause Mortality
Description: The total number of hospitalisations for myocardial infarction (MI) or all-cause mortality is reported using the adjusted event rate.
  The adjusted event rate is based on a negative binomial model adjusted for factors for treatment and type-2 diabetes at baseline, geographical region, age at baseline, estimated glomerular filtration rate at baseline, left ventricular ejection fraction at baseline, persistent or permanent atrial fibrillation at baseline, prior myocardial infarction at baseline, peripheral artery disease at baseline and smoking at baseline as covariates. The log(observation time) was used as an offset variable.
Time Frame: as for outcome 1
Population: Randomised set (RS): All randomised patients, whether treated or not.
Measure: Number (95% Confidence Interval); unit: Events/100 patient-years at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3262 | 3260
Events/100 patient-years at risk | 6.27 [5.19 to 7.58] | 6.66 [5.49 to 8.08]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.6311, Negative binomial regression; Adjusted event rate ratio = 1.06, 95% CI 2-sided [0.83 to 1.35] — Empagliflozin vs. Placebo

6. Secondary Outcome: Time to Cardiovascular (CV) Mortality
Description: The time to cardiovascular (CV) mortality is reported as the incidence rate of cardiovascular (CV) mortality, including deaths of unknown cause.
  The incidence rate was calculated as: the number of patients with a cardiovascular death event by treatment group during time at risk divided by the total time patients were at risk in that treatment group multiplied by 100 (per 100 Pt-years, Pt as abbreviation of patient).
Time Frame: as for outcome 1
Population: Randomised set (RS): All randomised patients, whether treated or not.
Measure: Number (95% Confidence Interval); unit: Pt with events/100 pt-years at risk
Arm/Group | Placebo | Empagliflozin 10 mg
Number analyzed (Participants) | 3262 | 3260
Pt with events/100 pt-years at risk | 2.76 [2.31 to 3.25] | 2.78 [2.33 to 3.28]
Statistical Analysis 1: Comparison: Placebo vs Empagliflozin 10 mg; Test type: Other — The statistical analysis was performed using a Cox proportional hazards model with treatment, type-2 diabetes at baseline, geographical region, age at baseline, estimated glomerular filtration rate at baseline, left ventricular ejection fraction at baseline, persistent or permanent atrial fibrillation at baseline, prior myocardial infarction at baseline, peripheral artery disease at baseline and smoking at baseline as covariates; p = 0.8124, Regression, Cox; Hazard Ratio (HR) = 1.03, 95% CI [0.81 to 1.31] — Empagliflozin vs. Placebo

ADVERSE EVENTS:
Time Frame: All-cause mortality - From first drug administration until individual day of trial completion. Up to 1004 days. Adverse event reporting - From first study drug administration to last study drug administration plus 7 days (residual effect period). Up to 1004 days.
Description: All-cause mortality- Randomised set: All randomised patients, whether treated or not.
  Adverse event reporting - Treated set: all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment.
Arm/Group | Placebo | Empagliflozin 10 mg
All-Cause Mortality (participants affected / at risk) | 178/3262 | 169/3260
Serious Adverse Events (participants affected / at risk) | 798/3229 | 765/3234
Other Adverse Events (participants affected / at risk) | 0/3229 | 0/3234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=3229) | Empagliflozin 10 mg (N=3234)
Anaemia (Blood and lymphatic system disorders) | 11 | 9
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 5
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 28 | 30
Angina unstable (Cardiac disorders) | 54 | 52
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 3
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arrhythmic storm (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 17 | 18
Atrial flutter (Cardiac disorders) | 3 | 6
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 5 | 3
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 5 | 2
Cardiac aneurysm (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 17 | 11
Cardiac failure (Cardiac disorders) | 230 | 159
Cardiac perforation (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 3 | 2
Cardiac ventricular disorder (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 4 | 11
Cardio-respiratory arrest (Cardiac disorders) | 5 | 6
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Chronic coronary syndrome (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 14 | 14
Coronary artery dissection (Cardiac disorders) | 2 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 2
Coronary artery stenosis (Cardiac disorders) | 4 | 4
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Dilated cardiomyopathy (Cardiac disorders) | 0 | 1
Dressler's syndrome (Cardiac disorders) | 0 | 3
Interventricular septum rupture (Cardiac disorders) | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 3 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 2
Microvascular coronary artery disease (Cardiac disorders) | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 94 | 110
Myocardial injury (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 6 | 0
Myocardial rupture (Cardiac disorders) | 1 | 1
Nodal rhythm (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Papillary muscle rupture (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 3 | 4
Pericardial haemorrhage (Cardiac disorders) | 1 | 1
Pericarditis (Cardiac disorders) | 4 | 3
Postinfarction angina (Cardiac disorders) | 0 | 2
Prinzmetal angina (Cardiac disorders) | 0 | 1
Sinus arrest (Cardiac disorders) | 1 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 3 | 1
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 3
Tachycardia (Cardiac disorders) | 0 | 1
Ventricle rupture (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 3
Ventricular extrasystoles (Cardiac disorders) | 2 | 2
Ventricular fibrillation (Cardiac disorders) | 3 | 2
Ventricular flutter (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 22 | 18
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Buried penis syndrome (Congenital, familial and genetic disorders) | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 3
Diabetic retinopathy (Eye disorders) | 0 | 1
Macular degeneration (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal artery embolism (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 2
Retinal infarction (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Duodenal polyp (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 22 | 28
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 3
Intestinal angina (Gastrointestinal disorders) | 0 | 1
Intestinal metaplasia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 3
Mechanical ileus (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Oronasal fistula (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 3
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1
Pelvic floor hernia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Volvulus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 4 | 0
Cardiac death (General disorders) | 1 | 3
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 12 | 9
Death (General disorders) | 21 | 21
Gait disturbance (General disorders) | 1 | 1
Implant site haematoma (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 27 | 28
Physical deconditioning (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 4
Sudden cardiac death (General disorders) | 7 | 9
Sudden death (General disorders) | 12 | 11
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Vascular stent stenosis (General disorders) | 2 | 2
Vascular stent thrombosis (General disorders) | 3 | 3
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 2 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 2 | 0
Haemorrhagic cholecystitis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 6
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 2
Appendicitis (Infections and infestations) | 2 | 5
Arthritis bacterial (Infections and infestations) | 2 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 25 | 20
COVID-19 pneumonia (Infections and infestations) | 10 | 14
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 1
Complicated appendicitis (Infections and infestations) | 1 | 0
Coronavirus infection (Infections and infestations) | 1 | 0
Coronavirus pneumonia (Infections and infestations) | 1 | 1
Dental fistula (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 3
Endocarditis (Infections and infestations) | 1 | 1
Endotoxic shock (Infections and infestations) | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 1
Gastroenteritis aeromonas (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected fistula (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 2 | 0
Joint abscess (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Norovirus infection (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 1
Perineal infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 30 | 31
Postoperative wound infection (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 8 | 9
SARS-CoV-2 viraemia (Infections and infestations) | 1 | 0
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 6 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 9
Urosepsis (Infections and infestations) | 0 | 2
Vestibular neuronitis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 1 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Aortic injury (Injury, poisoning and procedural complications) | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 3
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 2 | 0
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 2
Femur fracture (Injury, poisoning and procedural complications) | 4 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Neck injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 9
Post procedural stroke (Injury, poisoning and procedural complications) | 0 | 1
Postoperative delirium (Injury, poisoning and procedural complications) | 1 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0
Strangulated incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 2
Surgical procedure repeated (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood pressure increased (Investigations) | 1 | 1
Clostridium test positive (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Stress echocardiogram abnormal (Investigations) | 1 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 6 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Oligoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Lung squamous cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mucoepidermoid carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Rectosigmoid cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 4
Carotid artery thrombosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral hypoperfusion (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 4 | 6
Cerebral ischaemia (Nervous system disorders) | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 8 | 8
Cortical laminar necrosis (Nervous system disorders) | 0 | 1
Dementia (Nervous system disorders) | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 4
Epilepsy (Nervous system disorders) | 3 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Intracranial mass (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 11 | 7
Lacunar infarction (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Post-traumatic epilepsy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 3 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Ruptured cerebral aneurysm (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 2
Status epilepticus (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 2
Syncope (Nervous system disorders) | 19 | 16
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Tremor (Nervous system disorders) | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1
Vertebral artery occlusion (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Vertebrobasilar stroke (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 0 | 1
Mania (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 43 | 27
Bladder disorder (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 4 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 10 | 5
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 1
Nephropathy toxic (Renal and urinary disorders) | 9 | 6
Oliguria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 2
Renal haematoma (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 2 | 1
Renal infarct (Renal and urinary disorders) | 0 | 2
Ureterolithiasis (Renal and urinary disorders) | 2 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 4 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 2
Penile scarring (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Physical assault (Social circumstances) | 1 | 0
Tobacco user (Social circumstances) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 1 | 0
Acute aortic syndrome (Vascular disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 3
Aortic stenosis (Vascular disorders) | 1 | 1
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Blood pressure inadequately controlled (Vascular disorders) | 1 | 1
Circulatory collapse (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2
Extremity necrosis (Vascular disorders) | 1 | 3
Femoral artery embolism (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 3 | 3
Hypertensive crisis (Vascular disorders) | 5 | 7
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 7 | 8
Hypovolaemic shock (Vascular disorders) | 1 | 1
Iliac artery arteriosclerosis (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2
Peripheral artery occlusion (Vascular disorders) | 1 | 2
Peripheral embolism (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 3
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Subclavian vein stenosis (Vascular disorders) | 1 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 1
Vasoconstriction (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/74/NCT04509674/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/74/NCT04509674/SAP_001.pdf